CLINICAL TRIAL: NCT05887323
Title: Left Bundle Branch Area Pacing (LBBAP) Data Collection Registry
Brief Title: LBBAP Data Collection Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10474
Record Dates: First submitted 2023-04-27; First posted 2023-06-02 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Bradycardia; Sinus Node Dysfunction; Heart Block; Syncope; Cardiomyopathies; Heart Failure
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome; Heart Block; Syncope; Cardiomyopathies; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Left Bundle Branch Area Implant: Data included in this LBBAP data collection registry will be from subjects followed for 6 months (± 3 months) after attempted implant of LBBAP location. Data will be collected from previously occurring visits at pre-implant (baseline, required), implant (required), 6 months (±3 months, required), and 12 months (-2, +4months, optional).
  Interventions: Device: Implantation of the Tendril 2088 lead in the LBBA

INTERVENTIONS:
Device: Implantation of the Tendril 2088 lead in the LBBA — Conduction system pacing is achieved by delivering a pacing stimulus to the Left Bundle Branch area of the heart with Abbott's Tendril 2088 lead.

SUMMARY:
The purpose of this registry is to evaluate the safety and effectiveness of LBBA pacing/sensing in patients already implanted with the Tendril STS 2088 lead.

DETAILED DESCRIPTION:
This registry is a retrospective, observational, non-controlled chart review conducted to support an indication expansion of the Tendril STS 2088 lead to include pacing/sensing in the left bundle branch area.

Data from a minimum of 220 attempted subjects will be included in order to have 190 evaluable subjects in this registry. The chart review will be conducted at up to 20 participating centers worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a de novo attempted implant of the TendrilTM STS 2088 lead in the Left Bundle Branch Area on or before January 31, 2023 and subject's medical records contain data through at least 6 months (+/- 3 months) after LBBAP implant attempt
2. Subject is ≥ 18 years of age or the legal age, whichever age is greater
3. For sites where the governing IRB/EC has not granted a waiver of informed consent, subject has either been informed of the nature of the clinical investigation using a privacy notice or has provided a signed written informed consent, as approved by the IRB/EC (Note: This inclusion criterion is not applicable for sites where the governing IRB/EC or applicable regulation has granted a waiver of patient consent)

Exclusion Criteria:

1. Subject was enrolled in another clinical trial during this data collection period that might impact the outcomes of the present registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an attempted LBBA implant with Abbott's Tendril 2088 lead
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwangdeok Lee, Study Director — Abbott
Locations (11):
- United States (5):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Eisenhower Medical Center, Rancho Mirage, California
  - Cardiology Consultants - Baptist Campus, Pensacola, Florida
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Geisinger Medical Center, Danville, Pennsylvania
- Hopital d'adulte de la Timone, Marseille, Alpes, France
- India (2):
  - Medanta - The Medicity Hospital, Gūrgaon, NCT DLH
  - The Madras Medical Mission, Chennai, Tamil Nadu
- Ospedale S.Maria della Misericordia, Rovigo, Veneto, Italy
- Singapore (2):
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Left Bundle Branch Area Implant
Started | 221
Implant Attempt | 221
6-Month | 221
Completed | 221
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Left Bundle Branch Area Implant
Number analyzed (Participants) | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 34
  >=65 years | 186
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Singapore | 80
  United States | 78
  Italy | 5
  France | 25
  India | 33
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percentage] — Population: Left ventricular ejection fraction data were available only in 178 patients.
  percentage
    number analyzed (Participants) | 178
    (all) | 53.3 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint Evaluates Freedom From LBBAP Lead Related Serious Adverse Device Effects (SADEs).
Description: The primary safety endpoint evaluates a LBBAP lead related SADE rate which is an appropriate measure for safety and consistent with the primary safety endpoints used for evaluating performance of the transvenous right ventricular lead.
Time Frame: 6 months after the implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Left Bundle Branch Area Implant
Number analyzed (Participants) | 221
Participants | 220

2. Primary Outcome: The Primary Effectiveness Endpoint Evaluates the Composite Success Rate of Acceptable Capture Thresholds and Sense Amplitudes for LBBAP
Description: The primary effectiveness endpoint evaluates the ability to pace and sense when the TendrilTM STS 2088 lead is implanted in the LBBA. This analysis was performed on the successfully implanted population.
Time Frame: 6 months after the implantation
Population: This analysis was performed on the successfully implanted population.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Bundle Branch Area Implant
Number analyzed (Participants) | 201
Participants | 187

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Left Bundle Branch Area Implant
All-Cause Mortality (participants affected / at risk) | 5/221
Serious Adverse Events (participants affected / at risk) | 5/221
Other Adverse Events (participants affected / at risk) | 4/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Left Bundle Branch Area Implant (N=221)
Heart Failure (Cardiac disorders) | 3
Acute Decompensated Heart Failure (Cardiac disorders) | 1
Lead Dislodgement or Migration (Product Issues) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Left Bundle Branch Area Implant (N=221)
Developed Atrial Fibrillation with Atrial Lead (Cardiac disorders) | 1
Mechanical Bump to Right Bundle Branch Resulting in Complete Heart Block (Cardiac disorders) | 1
Bruising and Swelling at Insertion Site (General disorders) | 1
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are permitted to publish study-related results according to the local study contract and protocol. Draft publications or presentations must be provided to the Sponsor prior to any submission to determine if any confidential information is disclosed. Upon Sponsor request, the public disclosure may be delayed to enable the Sponsor to secure proprietary protection. The Sponsor shall not exercise editorial control over the proposed publication other than to correct technical accuracy.

DOCUMENTS (2):
  • Study Protocol (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT05887323/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT05887323/SAP_001.pdf